CLINICAL TRIAL: NCT03794128
Title: An Observational Feasibility Study for the Production of a Patient-Specific Neoantigen Cancer Vaccine and Screening Study for a Shared Neoantigen Cancer Vaccine in Patients With Advanced Cancer
Brief Title: A Study of Personalized Neoantigen Cancer Vaccines
Status: Completed | Type: Observational
Sponsor: Gritstone bio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GO-003
Record Dates: First submitted 2018-12-18; First posted 2019-01-04 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Non Small Cell Lung Cancer; Colorectal Cancer; Gastroesophageal Adenocarcinoma; Urothelial Carcinoma; Pancreatic Ductal Adenocarcinoma
Keywords: neoantigen cancer vaccine; personalized neoantigen cancer vaccine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Carcinoma, Transitional Cell | interventions — High-Throughput Nucleotide Sequencing; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * whole blood specimen, for HLA typing (all participants)
  * FFPE tumor material from a biopsy or resection, for sequencing to identify tumor-specific mutations (Group 1 participants only)
  * whole blood specimen, for sequencing of normal genome (Group 1 participants only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 - patient-specific neoantigen cancer vaccine production
  Interventions: Procedure: Blood collection for research (next-generation sequencing [NGS]); Procedure: Blood collection for research (HLA typing)
- 2 - shared neoantigen cancer vaccine screening
  Interventions: Procedure: Blood collection for research (HLA typing)

INTERVENTIONS:
Procedure: Blood collection for research (next-generation sequencing [NGS]) — Participants will have whole blood collected for next-generation sequencing (NGS).
  Groups: 1 - patient-specific neoantigen cancer vaccine production
Procedure: Blood collection for research (HLA typing) — Participants will have whole blood collected for HLA typing.

SUMMARY:
The purpose of this study is 1) to evaluate the feasibility of manufacturing a patient-specific neoantigen cancer vaccine, which involves predicting the patient's neoantigens and generating a vaccine that encodes the predicted neoantigens; and, 2) to identify and select patients who may be eligible for a shared neoantigen cancer vaccine where their tumor contains a specific shared mutation and who have the correct HLA allele capable of presenting the neoantigen derived from the tumor-specific mutation.

DETAILED DESCRIPTION:
Gritstone is developing two neoantigen-based cancer vaccines: the first is a patient-specific cancer vaccine that requires a manufacturing period for each patient and the second is an off-the-shelf cancer vaccine that targets shared neoantigens.

The process of generating a patient-specific neoantigen cancer vaccine involves multiple steps, including collection of patient tumor and blood specimens, performing next-generation sequencing (NGS), predicting the neoantigens to be included in the patient-specific vaccine, and the manufacture and release of the patient-specific vaccine. Gaining experience in managing the manufacturing process will provide important insights and experience regarding this process to be used in operationalizing future clinical trials.

Selecting patients who may be eligible to receive a shared neoantigen vaccine requires first identifying patients whose tumor possesses a neoantigen derived from an oncogenic mutation that is encoded by the vaccine, and then determining whether the patient expresses a matching HLA allele for antigen presentation.

Study participants will not receive any investigational treatment as part of this trial. Patients screened in this study may be able to enroll in a separate investigational treatment study sponsored by Gritstone Oncology, provided that the patient meets the specified eligibility criteria for that treatment study.

ELIGIBILITY:
Group 1 Inclusion Criteria:

* Provide a signed and dated informed consent form prior to initiation of study-specific procedures
* Patients with the indicated advanced or metastatic solid tumor as follows:

  1. NSCLC who have received ≤ 1 cycle of systemic treatment with cytotoxic, platinum-based chemotherapy (Note: patients with NSCLC who are receiving pembrolizumab monotherapy as first line systemic monotherapy are eligible)
  2. GEA who have received ≤ 1 cycle of systemic treatment with cytotoxic, platinum-based chemotherapy
  3. mUC who have received ≤ 1 cycle of systemic treatment with cytotoxic, platinum-based chemotherapy
  4. CRC-microsatellite stable (MSS) who have received ≤ 1 cycle of second line systemic therapy including a fluoropyrimidine and oxaliplatin or irinotecan (Note: patients receiving first-line systemic therapy are eligible)
* 18 years of age or older
* ECOG Performance Status 0 or 1
* Available FFPE tumor specimen for sequencing and neoantigen selection
* Measurable disease according to RECIST v1.1 Have adequate organ function, as measured by laboratory values (criteria listed in protocol)

Group 1 Exclusion Criteria:

* Tumors with genetic characteristics as follows:

  1. For NSCLC, patients with a known driver genomic alteration in EGFR, ALK, ROS1, RET, or TRK
  2. For CRC or GEA, patients with MSI disease
  3. For CRC, patients with a known BRAF mutation or patients with peritoneal carcinomatosis

Group 2 Inclusion Criteria:

* Provide a signed and dated informed consent form prior to initiation of study-specific procedures
* Patient's tumor possesses one of the mutations listed in the clinical study protocol, as determined per local institutional standard
* Patients with an advanced or metastatic solid tumor as follows:

  1. MSS-CRC who are currently receiving systemic treatment with a fluoropyrimidine and oxaliplatin or irinotecan that may include a VEGF or EGFR targeting therapy as their first-line or second-line therapy for metastatic disease
  2. NSCLC who are currently receiving systemic treatment with cytotoxic, platinum-based chemotherapy in combination with an anti-PD-(L)1 antibody
  3. PDA who are currently receiving systemic cytotoxic chemotherapy as their first-line therapy for metastatic disease

Group 2 Exclusion Criteria

* Patients with MSI disease
* Patients with NSCLC with a known driver genomic alteration in EGFR, ALK, ROS1, RET, or TRK

Complete inclusion and exclusion criteria are listed in the clinical study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Group 1 only: Presence of neoantigens sufficient to warrant patient-specific vaccine manufacture | At study enrollment
Group 1 only: Percentage of patients for whom patient-specific vaccine is successfully manufactured (defined as meeting release criteria) | Up to approximately 20 weeks
Group 2 only: Percentage of patients with at least one of the twenty specified shared mutations contained in the expression cassette and a matching HLA allele for neoantigen presentation | Up to approximately 2 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois
  - Columbia University Medical Center, Herbert Irving Comprehensive Cancer Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Tennessee Oncology, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia